CLINICAL TRIAL: NCT05780801
Title: Sentinel Cohort for the Response to Emerging Antimicrobial Resistance With Containment Microbiota Restoration Therapy Trial
Brief Title: Sentinel Cohort REACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Woodworth, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005467; U54CK000601 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-23 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Multi-Drug Resistant Organism
Keywords: Multi-Drug Resistant Pseudomonas; Clostridioides difficile; Carbapenem-resistant Enterobacteriaceae (CRE); Vancomycin-Resistant Enterococcus (VRE); Extended Spectrum Beta-Lactamase (ESBL)
MeSH Terms: interventions — Glycerol; Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Live microbiome therapeutic (Experimental): Live microbiome therapeutic prepared as Allogeneic Microbiota in Glycerol (10%) (AMG)
  Interventions: Drug: Allogeneic Microbiota in Glycerol (10%) (AMG)

INTERVENTIONS:
Drug: Allogeneic Microbiota in Glycerol (10%) (AMG) — Participants with positive MDRO cultures will receive MT instilled via a functional feeding tube when in place or rectal enema (when a functional feeding tube is not present) with the rate adjusted to the recipient's clinical status and infusion tolerance.
  Other Names: Stool from healthy donors in saline suspension with 10% glycerol by volume; Fecal Microbiota Transplant (FMT); Microbiome therapeutic

SUMMARY:
The purpose of this study is to better understand the efficacy and safety of microbiome therapies (MT) in patients with Multidrug Resistant Organism (MDRO) colonization who are admitted to Long Term Acute Care Hospitals (LTACH). This use of MT has been studied in other small studies to treat MDRO colonization, further study of the effect of MT on the transmission of MDRO to other patients is needed. This study will test the safety of the MT for this use in LTACH patients, and how well it works to help design larger studies.

Importance to the field: MDRO colonization increases the risk of subsequent infection and transmission to others, however, there are no approved therapies for decolonization or reduction of the burden of colonization with MDROs. MT like Allogeneic Microbiota in Glycerol (AMG) has been shown to have ~ 60-90% efficacy for decolonization and an acceptable safety profile but has not been studied in this population for this indication.

Study population: patients admitted to long-term care facilities (e.g. LTACHs and ventilator-capable skilled nursing facilities [vSNF]) found to be MDRO colonized during prevalence screening activities. The MT AMG will be delivered through an already existing feeding tube or into the rectum as an enema.

DETAILED DESCRIPTION:
This protocol describes an open-label sentinel cohort study of MT treatment of 10-20 participants who are admitted to an LTACH or vSNF and colonized by a target MDRO as detected by peri-rectal or stool culture. Safety data from this sentinel cohort were requested by the FDA in advance of a larger multi-center study called REACT. This study is conducted in two parts. In part 1 (under a linked IRB protocol), facilities undergo periodic point prevalence sampling for the qualitative detection of patient MDRO colonization with culture-based assays. In part 2 (the present protocol) all MDRO-positive patients at a participating facility will be offered MT for MDRO decolonization with safety and efficacy follow-up.

Bacterial isolates will be subjected to whole-genome sequencing. Swabs (e.g. peri-rectal/stool, inguinal) will be stored for metagenomic sequencing. Sequencing data are required to be shared in public repositories but sequencing reads that map to reference human genomes are removed, which should greatly reduce the risk of potential identifiability of human genetic content in these datasets.

ELIGIBILITY:
Inclusion Criteria:

* Be able to (or have an available Legal Authorized Representative who is able to) understand and be willing to sign a written informed consent document.
* Be at least 18 years old at the time of consent.
* Be able and willing to comply with all study protocol requirements, including being willing to receive MT through a feeding tube or as a retention enema.
* Be colonized with a target MDRO (CRE, VRE, ESBL, MDR Pseudomonas, and/or C. difficile) as detected by bacterial culture of stool or peri-rectal swab.
* Be willing to discontinue antibiotics, probiotics, other microbiota restoration therapies, and proton pump inhibitors (PPIs) at least one day prior to study Day 0 up to Day 28.
* The effects of the IP on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* If the potential participant is male and is sexually active with a partner of childbearing potential, the participant agrees to practice at least one effective method of birth control for the duration of the study.
* A negative urine human chorionic gonadotropin (hCG) testing on the day of FMT for women of childbearing potential (WOCBP), to proceed with FMT.

Exclusion Criteria:

* Be pregnant, breastfeeding, lactating, or planning a pregnancy during the study duration (through 4 weeks after the last dose of the investigational product (IP)), if women of childbearing potential (WOCBP).
* Have known uncontrolled intercurrent illness(es) such as, but not limited to: Symptomatic congestive heart failure, acute coronary syndrome, or cardiac arrhythmia, untreated in-situ colorectal cancer, toxic megacolon, ileus, positive stool studies without completion of treatment course (including ova and parasites, Salmonella spp, Shigella, Campylobacter, and other enteropathogens)
* Have any other intercurrent acute illness that in the opinion of the investigator will preclude the subject from entering the study.
* Be on systemic antibiotics for any reason other than treatment of recent MDRO infection or clear anticipated need for antibiotics during the follow-up period that cannot be rescheduled (e.g. fluoroquinolone prophylaxis for percutaneous nephrostomy tube exchange). Participants must complete the planned antibiotic course by study Day -1.
* Inability to discontinue proton-pump inhibitor therapy.
* Have a compromised immune system, defined as AIDS with clusters of differentiation 4 (CD4)+ T-cell count <200 and any detectable HIV viral load, absolute neutrophil count (ANC) <1,000 neutrophils / mL on the day of enrollment, active malignancy requiring intensive induction chemotherapy, radiotherapy, or biologic treatment within 2 months of enrollment or history of hematopoietic cell transplantation, either allogeneic or autologous in the last 1 year.
* Have a history of significant food allergy that led to anaphylaxis or hospitalization.
* Have a life expectancy of 24 weeks or less
* Have any condition that, in the opinion of the investigator, might interfere with study objectives or limit compliance with study requirements, including but not limited to: Known active intravenous drug or alcohol abuse, psychiatric illness, and/or social situation
* Participated in an investigational study that also meets one of the following criteria: has received an interventional agent (drug, device, or procedure) in the last 28 days or has enrolled in any other interventional study for MDROs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events by MT administration in a population with a high burden of comorbidities | Day 7
  Frequency of adverse events from MT administration up to 1 week.
Severity of adverse events caused by administration for MT in a population with a high burden of comorbidities | Day 7
  Severity of adverse events is to be graded as mild, moderate or severe, form the time of MT administration up to 1 week.
Frequency of adverse events by MT administration in a population with a high burden of comorbidities | Day 0 up to 196 days
  All adverse events will be documented from MT administration up to day 28 + 6 months.
Severity of adverse events caused by administration for MT in a population with a high burden of comorbidities | Day 0 up to 196 days
  The severity of adverse events will be documented from MT administration up to day 28 + 6 months.

SECONDARY OUTCOMES:
MT MDRO decolonization efficacy | Day 14
  MT MDRO decolonization efficacy will be estimated by the proportion of MT-recipient stool cultures positive for any target MDRO

CONTACTS AND LOCATIONS:
Overall Officials: Michael Woodworth, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Emory Long-Term Acute Care, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share the Cultured isolate MDRO category for study inclusion, the 7-day safety data (frequency & severity of adverse events), MDRO culture results at 4 weeks, and all the genomic/metagenomic data analyzed in any presented or published results.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared at the time of publication.
Access Criteria: The investigators will share fully deidentified data and sequencing data which will be uploaded to a repository (e.g. Dataverse or similar) and access will not be restricted.

REFERENCES:
- [Derived] Woodworth MH, Babiker A, Prakash-Asrani R, Mehta CC, Steed DB, Ashley A, Koundakjian D, Acharya A, Grooms L, Bower CW, Suchindran DR, Trehan T, Halpin AL, Spalding Walters M, Reddy SC, Samore MH, Roghmann MC, Hayden MK, Van Riel J, Burd EM, Lohsen S, Satola SW, Fridkin SK. Microbiota Transplantation Among Patients Receiving Long-Term Care: The Sentinel REACT Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2522740. doi: 10.1001/jamanetworkopen.2025.22740. PMID 40705333

DOCUMENTS (1):
  • Informed Consent Form (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT05780801/ICF_000.pdf